CLINICAL TRIAL: NCT03503799
Title: Prospective Assessment of Disease Progression in Primary Breast Cancer Patients Undergoing EndoPredict® Gene Expression Testing - a Care Research Study
Brief Title: Reaching for Evidence-baSed Chemotherapy Use in Endocrine Sensitive Breast Cancer
Acronym: RESCUE
Status: Active, not recruiting | Type: Observational
Sponsor: North Eastern German Society of Gynaecological Oncology (Other)
Collaborators: Center for Clinical Trials Philipps University Marburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: NOGGO B3
Record Dates: First submitted 2018-03-19; First posted 2018-04-20 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Primary Invasive Breast Cancer; Estrogen Receptor Positive Tumor; Human Epidermal Growth Factor Receptor 2 Negative Tumor
Keywords: breast cancer; EndoPredict®; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational Group: Patients with primary invasive breast cancer, Stage I/II; ER positive, HER2 (human epidermal growth factor receptor 2) negative, N0-N1, T1-T3, tested with EndoPredict®, age over 18 years, informed consent
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Visit 1 Informed consent Medical history Demographics Result of EndoPredict® Test Status of menopause Disease status Tumor board decision Planned anti-tumor-therapy
  Visit 2, 1 year after inclusion This visit will be documented at the study site Status of menopause Disease status Anti-tumor therapy Survival
  Following visits For these visits, patients will be asked directly through the Center for Clinical Trials of the Philipps-University Marburg (KKS Marburg) via phone.
  Status of Menopause Disease status Anti-tumor therapy Survival
  Treatment after end of the study The patient will be treated during and after end of study by physician's choice.

SUMMARY:
Systematic assessment of survival data of patients who have been tested with EndoPredict®; prospective proof that patients with low risk classification by EndoPredict® (EPclin) can safely forgo chemotherapy and be treated with endocrine therapy alone.

DETAILED DESCRIPTION:
The goal of the study is to receive current and comprehensive information about the diseasefree (remote metastasis free and recurrence free) interval of EndoPredict® low risk patients.

The study is organized and managed by the NOGGO e.V. (North Eastern German Society of Gynaecological Oncology e.V.) study coordination office under the existing and efficient infrastructure. All patients who receive gene expression analysis with EndoPredict® and satisfy the remaining inclusion / exclusion criteria may participate in the study. Data collection is prospective and non-interventional. The recruitment of the required patients is expected to take a maximum of 36 months .

It must be emphasized that the study is data collection only and not an interventional study. This means that the choice and implementation of the therapy as well as the treatment assessments and frequency during and after the treatment can only be determined by the Investigator.

The decision to participate in the study is independent of the patient´s therapy within the framework of a study. Patient data will be recorded at the time of inclusion and once a year thereafter. Patient follow-up will be by phone from the second year onward.

Primary objective is to show that female patients who have been tested as "low risk" by EPclin and have been treated with endocrine therapy only for at least 5 years have a 10-year DMFS rate > 90% (lower boundary of the one-sided 95% confidence interval).

Secondary objectives comprise the evaluation of DMFS (distant metastasis free survival) , DFS (disease free survival) and OS (overall survival) rates at different time points and for different groups. Assessment of the given chemotherapy regimens and the given endocrine therapy will be performed and the proportions of patients will be determined with respect to the received treatment and its duration in different groups. Furthermore, the proportion of patients in whom the tumor board recommendation follows the EndoPredict® result and the proportion of patients actually treated according to EndoPredict® result will be determined.

The association between outcome and treatment, EPclin, EP, and classical prognostic factors will be investigated in different groups of patients. The correlation and concordance between EPclin calculations derived from biopsies and surgical specimens will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent
2. Tested with EndoPredict within the previous 6 months before inclusion
3. Age ≥ 18 years
4. Patients with primary invasive breast cancer, Stage I/II
5. ER-positive
6. HER2-negative
7. N0 or N1 (1-3 positive lymph nodes)
8. T1 - T3

Exclusion Criteria:

1. Inflammatory breast cancer
2. Bilateral breast cancer
3. Breast cancer in the last 10 years
4. Other invasive malignancies in the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary stage I or Ii breast cancer who met all inclusin and no exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1191 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2032-10-01 (Estimated); Study Completion 2032-10-01 (Estimated)

PRIMARY OUTCOMES:
Distant metastasis free survival | 10 years
  To show that female patients who have been tested as "low risk" by EndoPredict® (EPclin) and have been treated with endocrine therapy only for at least 5 years have a 10-year distant metastasis-free survival (DMFS) > 90 % (lower boundary of the one-sided 95 % confidence interval)

SECONDARY OUTCOMES:
DMFS "low risk" | 3, 5 and 10 years
  Assessment of DMFS of patients with EPclin "low risk" (or EP "low risk" [EP score <5] if EPclin cannot be calculated after surgery in the neoadjuvant setting) (in all patients, in the relevant target group and separately in men and women and in pre- and postmenopausal women with regard to treatment).
DFS "low risk" | 3, 5 and 10 years
  Assessment of DFS of patients with EPclin "low risk" (or EP "low risk" [EP score <5] if EPclin cannot be calculated after surgery in the neoadjuvant setting) (in all patients, in the relevant target group and separately in men and women and in pre- and postmenopausal women with regard to treatment).
OS "low risk" | 3, 5 and 10 years
  Assessment of OS of patients with EPclin "low risk" (or EP "low risk" [EP score <5] if EPclin cannot be calculated after surgery in the neoadjuvant setting) (in all patients, in the relevant target group and separately in men and women and in pre- and postmenopausal women with regard to treatment).
DMFS "high risk" | 3, 5 and 10 years
  Assessment of DMFS of patients with EPclin "high risk" in all patients and separated in men and women as well as pre- and postmenopausal women with regard to treatment).
DFS "high risk" | 3, 5 and 10 years
  Assessment of DFS of patients with EPclin "high risk" in all patients and separated in men and women as well as pre- and postmenopausal women with regard to treatment).
OS "high risk" | 3, 5 and 10 years
  Assessment of OS of patients with EPclin "high risk" in all patients and separated in men and women as well as pre- and postmenopausal women with regard to treatment).
DMFS "high risk + low risk" | 3, 5 and 10 years
  DMFS for patients who have / have not been treated according to EPclin/ EP result (all patients and subgroup analyses as specified in secondary objectives 1 and 2).
DFS "high risk + low risk" | 3, 5 and 10 years
  DFS for patients who have / have not been treated according to EPclin/ EP result (all patients and subgroup analyses as specified in secondary objectives 1 and 2).
OS "high risk + low risk" | 3, 5 and 10 years
  OS for patients who have / have not been treated according to EPclin/ EP result (all patients and subgroup analyses as specified in secondary objectives 1 and 2).
Portion of patients tumor board follows the EndoPredict® result | 1 year
  Assessment of the proportion of patients in whom the tumor board follows the EndoPredict® result in regard to treatment recommendation (in all patients and separately for men and women).
Portion of patient treated according EndoPredict® result | 1 year
  Assessment of the proportion of patients who were actually treated according to the EndoPredict® result (in all patients and separately for men and women).
Prognostic Performance of classical prognostic factors compared to EndoPredict® | 3, 5 and 10 years
  Assessment of the classical prognostic factors tumor size, nodal status, grading, quantitative estrogen receptor, quantitative progesterone receptor and quantitative Ki67 and evaluation of their prognostic performance compared to EPclin and EP in univariate and multivariate analyses of DMFS, DFS, OS (in all patients, separately for men and women, only in patients who have been treated according to the EndoPredict® result).
DMFS "low risk vs. high risk" | 3, 5 and 10 years
  Assessment of DMFS of patients with low risk vs. high risk as defined by national (German S3) and international (St. Gallen Consensus) guidelines based on IHC (immunohistochemistry)-classification.
DFS "low risk vs. high risk" | 3, 5 and 10 years
  Assessment of DFS of patients with low risk vs. high risk as defined by national (German S3) and international (St. Gallen Consensus) guidelines based on IHC-classification.
OS "low risk vs. high risk" | 3, 5 and 10 years
  Assessment of OS of patients with low risk vs. high risk as defined by national (German S3) and international (St. Gallen Consensus) guidelines based on IHC-classification.
DMFS of patient proportion of EPclin low and high risk patients in Ki67 low, intermediate and high tumors | 3, 5 and 10 years
  Assessment of proportion of EPclin low and high risk patients in Ki67 low, intermediate and high tumors, respectively, and stratified analysis of DMFS of patients with ki67-values low (≤ 10%)/ intermediate (11-24%)/ high (≥ 25%) and EPclin low risk vs high risk.
DFS of patient proportion of EPclin low and high risk patients in Ki67 low, intermediate and high tumors | 3, 5 and 10 years
  Assessment of proportion of EPclin low and high risk patients in Ki67 low, intermediate and high tumors, respectively, and stratified analysis of DFS of patients with ki67-values low (≤ 10%)/ intermediate (11-24%)/ high (≥ 25%) and EPclin low risk vs high risk.
OS of patient proportion of EPclin low and high risk patients in Ki67 low, intermediate and high tumors | 3, 5 and 10 years
  Assessment of proportion of EPclin low and high risk patients in Ki67 low, intermediate and high tumors, respectively, and stratified analysis of OS of patients with ki67-values low (≤ 10%)/ intermediate (11-24%)/ high (≥ 25%) and EPclin low risk vs high risk.
DMFS "low risk vs. high risk" who have /have not been treated according to the S3 and St. Gallen guidelines | 3, 5 and 10 years
  Assessment of DMFS after 3, 5 and 10 years of patients with low risk vs. high risk as defined by national (German S3) and international (St. Gallen Consensus) guidelines based on IHC-classification.
DFS "low risk vs. high risk" who have /have not been treated according to the S3 and St. Gallen guidelines | 3, 5 and 10 years
  Assessment of DFS of patients with low risk vs. high risk as defined by national (German S3) and international (St. Gallen Consensus) guidelines based on IHC-classification.
OS "low risk vs. high risk" who have /have not been treated according to the S3 and St. Gallen guidelines | 3, 5 and 10 years
  Assessment of OS of patients with low risk vs. high risk as defined by national (German S3) and international (St. Gallen Consensus) guidelines based on IHC-classification.
Chemotherapy regimens | 1 year
  Description of the given chemotherapy regimens (in all patients and separately for men and women).
Given endocrine therapy | 10 years
  Description of the given endocrine therapy (in all patients and separately for men and women).
Duration of endocrine therapy | 10 years
  Duration of the endocrine therapy (in all patients and separately for men and women).
Proportion of patients with prolonged endocrine therapy | 10 years
  Proportion of patients with EPclin "low risk" and "high risk" respectively who received an extended (> 5 years) endocrine therapy in all patients and separately for men and women).
DMFS for patients with 5 years of endocrine therapy vs. extended endocrine therapy | 10 years
  Assessment of DMFS according to EPclin / EP risk class for patients who have received an endocrine therapy for 5 years vs. patients who received an extended endocrine therapy (> 5 years).
DFS for patients with 5 years of endocrine therapy vs. extended endocrine therapy | 10 years
  Assessment of DFS according to EPclin / EP risk class for patients who have received an endocrine therapy for 5 years vs. patients who received an extended endocrine therapy (> 5 years).
OS for patients with 5 years of endocrine therapy vs. extended endocrine therapy | 10 years
  Assessment of OS according to EPclin / EP risk class for patients who have received an endocrine therapy for 5 years vs. patients who received an extended endocrine therapy (> 5 years).
Correlation ( pT- and pN data vs. ciT and ciN-data) | 1 year
  Assessment of the correlation between EPclin, that has been calculated with pT- (pathological tumor size) and pN (pathological nodal status) data and the EPclin based on ciT (clinical/ imaging tumor size) and ciN (clinical/imaging nodal status)-data (in all patients and separately for men and women).
Concordance ( pT- and pN data vs. ciT and ciN-data) | 1 year
  Assessment of the concordance between EPclin, that has been calculated with pT- and pN data and the EPclin based on ciT and ciN-data (in all patients and separately for men and women).

CONTACTS AND LOCATIONS:
Overall Officials: Marion Kiechle, Prof. Dr., Principal Investigator — TU München (TUM) Lehrstuhl für Gynäkologie und Geburtshilfe
Locations (40):
- Germany (37):
  - Frauenklinik der Technischen Universität München, München, Bavaria
  - Vivantes Klinikum am Urban, Berlin, State of Berlin
  - ANregiomed Ansbach, Ansbach
  - DRK Kliniken Köpenick, Berlin
  - MVZ Hellersdorf - Zweigstelle Biesdorf, Berlin
  - Park-Klinik Weißensee, Berlin
  - Helios Klinikum Berlin Buch, Berlin
  - Klinikum Bremerhaven Reinkenheide, Bremerhaven
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Krankenhaus St. Joseph Stift Dresden GmbH, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Evangelisches Krankenhaus, Düsseldorf
  - Kreisklinik Ebersberg, Ebersberg
  - Klinikum Erding, Erding
  - Praxis Dr. Heinrich, Fürstenwalde
  - Krankenhaus St. Elisabeth und St. Barbara, Halle
  - Krankenhaus Jerusalem, Hamburg
  - Asklepios Klinik Barmbek, Hamburg
  - Mathilden Hospital, Herford
  - Frauenärzte am Bahnhofsplatz, Hildesheim
  - Universitätsklinikum Jena, Jena
  - Gemeinschaftsklinikum Mittelrhein gGmbH Kemperhof, Koblenz
  - VK & K Studien GbR, Landshut
  - Krankenhaus St. Marienstift, Magdeburg
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Klinikum Fichtelgebirge, Marktredwitz
  - Charité - Universitätsmedizin Berlin, Mitte
  - Gemeinschaftspraxis Gynäkologie Arabella, München
  - Oberhavel Kliniken GmbH, Oranienburg
  - Regioklinik Pinneberg, Pinneberg
  - Ernst von Bergmann Klinikum, Potsdam
  - Universitätsklinikum Regensburg, Regensburg
  - RoMed Klinikum Rosenheim, Rosenheim
  - Klinikum Traunstein, Traunstein
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Harzklinikum Dorothea Christiane Erxleben, Wernigerode
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Switzerland (3):
  - Brustzentrum Bern Lindenhofgruppe, Bern
  - Luzerner Kantonsspital, Lucerne
  - Spital Zollikerberg, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Georgia Dental Service Corporation opens offices, signs contracts. J Ga Dent Assoc. 1968 Jul;42(1):12-4. No abstract available. PMID 5241904
- [Background] Cobain EF, Hayes DF. Indications for prognostic gene expression profiling in early breast cancer. Curr Treat Options Oncol. 2015 May;16(5):23. doi: 10.1007/s11864-015-0340-x. PMID 25929335
- [Background] Kim OH. Radionuclide detection and differential diagnosis of left-to-right cardiac shunts by analysis of time-activity curves. Osaka City Med J. 1986 Dec;32(2):65-88. No abstract available. PMID 3306560
- [Background] Denkert C, Pfitzner BM, Heppner BI, Dietel M. [Molecular pathology for breast cancer: Importance of the gene expression profile]. Pathologe. 2015 Mar;36(2):145-53. doi: 10.1007/s00292-015-0009-z. German. PMID 25836324
- [Background] Dubsky P, Brase JC, Jakesz R, Rudas M, Singer CF, Greil R, Dietze O, Luisser I, Klug E, Sedivy R, Bachner M, Mayr D, Schmidt M, Gehrmann MC, Petry C, Weber KE, Fisch K, Kronenwett R, Gnant M, Filipits M; Austrian Breast and Colorectal Cancer Study Group (ABCSG). The EndoPredict score provides prognostic information on late distant metastases in ER+/HER2- breast cancer patients. Br J Cancer. 2013 Dec 10;109(12):2959-64. doi: 10.1038/bjc.2013.671. Epub 2013 Oct 24. PMID 24157828
- [Background] Dubsky P, Filipits M, Jakesz R, Rudas M, Singer CF, Greil R, Dietze O, Luisser I, Klug E, Sedivy R, Bachner M, Mayr D, Schmidt M, Gehrmann MC, Petry C, Weber KE, Kronenwett R, Brase JC, Gnant M; Austrian Breast and Colorectal Cancer Study Group (ABCSG). EndoPredict improves the prognostic classification derived from common clinical guidelines in ER-positive, HER2-negative early breast cancer. Ann Oncol. 2013 Mar;24(3):640-7. doi: 10.1093/annonc/mds334. Epub 2012 Oct 3. PMID 23035151
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] Ettl J, Klein E, Hapfelmeier A, Grosse Lackmann K, Paepke S, Petry C, Specht K, Wolff L, Hofler H, Kiechle M. Decision impact and feasibility of different ASCO-recommended biomarkers in early breast cancer: Prospective comparison of molecular marker EndoPredict and protein marker uPA/PAI-1. PLoS One. 2017 Sep 6;12(9):e0183917. doi: 10.1371/journal.pone.0183917. eCollection 2017. PMID 28877230
- [Background] Filipits M, Rudas M, Jakesz R, Dubsky P, Fitzal F, Singer CF, Dietze O, Greil R, Jelen A, Sevelda P, Freibauer C, Muller V, Janicke F, Schmidt M, Kolbl H, Rody A, Kaufmann M, Schroth W, Brauch H, Schwab M, Fritz P, Weber KE, Feder IS, Hennig G, Kronenwett R, Gehrmann M, Gnant M; EP Investigators. A new molecular predictor of distant recurrence in ER-positive, HER2-negative breast cancer adds independent information to conventional clinical risk factors. Clin Cancer Res. 2011 Sep 15;17(18):6012-20. doi: 10.1158/1078-0432.CCR-11-0926. Epub 2011 Aug 1. PMID 21807638
- [Background] Fitzal F, Filipits M, Rudas M, Greil R, Dietze O, Samonigg H, Lax S, Herz W, Dubsky P, Bartsch R, Kronenwett R, Gnant M. The genomic expression test EndoPredict is a prognostic tool for identifying risk of local recurrence in postmenopausal endocrine receptor-positive, her2neu-negative breast cancer patients randomised within the prospective ABCSG 8 trial. Br J Cancer. 2015 Apr 14;112(8):1405-10. doi: 10.1038/bjc.2015.98. Epub 2015 Mar 24. PMID 25867274
- [Background] Kronenwett R, Bohmann K, Prinzler J, Sinn BV, Haufe F, Roth C, Averdick M, Ropers T, Windbergs C, Brase JC, Weber KE, Fisch K, Muller BM, Schmidt M, Filipits M, Dubsky P, Petry C, Dietel M, Denkert C. Decentral gene expression analysis: analytical validation of the Endopredict genomic multianalyte breast cancer prognosis test. BMC Cancer. 2012 Oct 5;12:456. doi: 10.1186/1471-2407-12-456. PMID 23039280
- [Background] Martin M, Brase JC, Calvo L, Krappmann K, Ruiz-Borrego M, Fisch K, Ruiz A, Weber KE, Munarriz B, Petry C, Rodriguez CA, Kronenwett R, Crespo C, Alba E, Carrasco E, Casas M, Caballero R, Rodriguez-Lescure A. Clinical validation of the EndoPredict test in node-positive, chemotherapy-treated ER+/HER2- breast cancer patients: results from the GEICAM 9906 trial. Breast Cancer Res. 2014 Apr 12;16(2):R38. doi: 10.1186/bcr3642. PMID 24725534
- [Background] Muller BM, Brase JC, Haufe F, Weber KE, Budzies J, Petry C, Prinzler J, Kronenwett R, Dietel M, Denkert C. Comparison of the RNA-based EndoPredict multigene test between core biopsies and corresponding surgical breast cancer sections. J Clin Pathol. 2012 Jul;65(7):660-2. doi: 10.1136/jclinpath-2012-200716. Epub 2012 Mar 23. PMID 22447922
- [Background] Muller BM, Keil E, Lehmann A, Winzer KJ, Richter-Ehrenstein C, Prinzler J, Bangemann N, Reles A, Stadie S, Schoenegg W, Eucker J, Schmidt M, Lippek F, Johrens K, Pahl S, Sinn BV, Budczies J, Dietel M, Denkert C. The EndoPredict Gene-Expression Assay in Clinical Practice - Performance and Impact on Clinical Decisions. PLoS One. 2013 Jun 27;8(6):e68252. doi: 10.1371/journal.pone.0068252. Print 2013. PMID 23826382
- [Background] Poremba C, Uhlendorff J, Pfitzner BM, Hennig G, Bohmann K, Bojar H, Krenn V, Brase JC, Haufe F, Averdick M, Dietel M, Kronenwett R, Denkert C. Preanalytical variables and performance of diagnostic RNA-based gene expression analysis in breast cancer. Virchows Arch. 2014 Oct;465(4):409-17. doi: 10.1007/s00428-014-1652-0. Epub 2014 Sep 14. PMID 25218890